CLINICAL TRIAL: NCT00883480
Title: Tratamiento Individualizado en función de Las Mutaciones en EGFR y Del Nivel de expresión de BRCA1 en Pacientes Con Adenocarcinoma de pulmón Avanzado
Brief Title: Individualized Treatment Based on Epidermal Growth Factor Receptor Mutations and Level of BRCA1 Expression in Advanced Adenocarcinoma
Acronym: SLAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spanish Lung Cancer Group (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SLAT
Record Dates: First submitted 2008-12-22; First posted 2009-04-17 (Estimated); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Cisplatin; Gemcitabine; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Experimental): The rest of the patients who do not carry the Factor Receptor mutation of Epidermal Growth will receive chemotherapy treatment individualized based on BRCA 1 m RNA levels. Function of these levels, three different subgroups of treatment: Subgroup A with low BRCA1 mRNA levels will receive treatment with gemcitabine / cisplatin Subgroup B with intermediate levels of BRCA1 mRNA: will receive treatment with docetaxel / cisplatin Subgroup C with high levels of BRCA1 mRNA: will receive treatment with docetaxel
  Interventions: Drug: Docetaxel; Drug: Cisplatin; Drug: Gemcitabine
- 1 (Experimental): The group of patients carrying EGFR mutation will receive treatment with Erlotinib, a selective oral Receptor tyrosine kinase inhibitor Epidermal Growth Factor
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 75 mg/day 1 x 4 cycles
  Other Names: Taxotere
  Arms: 2
Drug: Cisplatin — Docetaxel-Cisplatin 75 mg/day 1 x 4 cycles
  Other Names: Platinol
  Arms: 2
Drug: Gemcitabine — Cisplatin 75 mg/ day 1 x 4 cycles
  Gemcitabine 1250 mg/ day 1 and 8 x 4 cycles
  Other Names: Gemzar
  Arms: 2
Drug: Erlotinib — Erlotinib 150 mg/day x 21 days
  Other Names: Tarceva
  Arms: 1

SUMMARY:
This is a pharmacogenic, prospective, and multicenter study in patients with advanced lung adenocarcinoma.

DETAILED DESCRIPTION:
Pharmacogenomic study, prospective, multicenter. Individualized treatment based on EGFR mutations and level of BRCA1 expression in patients with advanced lung adenocarcinoma

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 years or more.
* Histologically confirmed diagnosis of non-small-cell lung carcinoma.(and indifferentiated and BAC histology).

  * Only patients with advanced disease, defined as stage IV or IIIB with/without pleural effusion, will be included.
  * Tumor sample available.
  * A measurable lesion, as defined by RECIST criteria.
  * Karnofsky score 60% or more (ECOG < 2).
  * Patients should not have received previous treatment with chemotherapy or other agents for disseminated disease. Chemotherapy is allowed if the initial diagnosis of the patient is limited disease and the patient has received adjuvant or neoadjuvant treatment.
* Patients with cerebral disease are permitted, without any time limitations after holocranial irradiation or complementary antiedema treatment.
* Patients with hepatical, renal and hematology normality values.
* Patients should sign an informed consent form before inclusion in the study that specifies that the clinical trial treatment entails consent for the analysis of biological samples of tumor and blood.
* Patients of childbearing age of either sex must use effective contraceptive methods (barrier methods or other birth control methods) before entering the study and while participating in the study.
* Patients must be available for clinical follow-up..

Exclusion Criteria:

* Patients who have received an investigational medicinal product in the 21 days before inclusion in the study or antiEGFR receptor agent.
* Severe comorbidity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2005-06; Primary Completion 2008-01 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Tumoral Response (RECIST criteria) | From date of end of experimental treatment until the date of last follow up, assessed up to 24 months]
  To evaluate the tumor response of the treatment as measured by investigator-assessed overall response rate according to RECIST v1.1.

SECONDARY OUTCOMES:
Overall Survival | From the date of randomization to the date of last follow up or death, assessed up to 24 months
  Time from randomization until death from any cause. Patients who have not died during the study will be tabulated on their last date of evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Rosell, MD, Study Chair — ICO-HOSPITAL GERMANS TRIAS I PUJOL
Locations (2):
- Spain (2):
  - Ico-Hospital Universitarios Germans Trias I Pujol, Badalona, Barcelona
  - Hospital Carlos Haya, Málaga

REFERENCES:
- [Derived] Rosell R, Perez-Roca L, Sanchez JJ, Cobo M, Moran T, Chaib I, Provencio M, Domine M, Sala MA, Jimenez U, Diz P, Barneto I, Macias JA, de Las Penas R, Catot S, Isla D, Sanchez JM, Ibeas R, Lopez-Vivanco G, Oramas J, Mendez P, Reguart N, Blanco R, Taron M. Customized treatment in non-small-cell lung cancer based on EGFR mutations and BRCA1 mRNA expression. PLoS One. 2009;4(5):e5133. doi: 10.1371/journal.pone.0005133. Epub 2009 May 5. PMID 19415121
- See also: Web page of the sponsor where users can find more information about Fundación GECP studies — http://www.gecp.org